CLINICAL TRIAL: NCT04825899
Title: A Non-interventional Study on the Relationship Between Gene Abnormalities and the Efficacy and Prognosis in Patients With Diffuse Large B-cell Lymphoma
Brief Title: Gene Abnormalities and Prognosis in Diffuse Large B-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junning Cao, MD, Chief Physician, Fudan University
Other Study IDs: gene abnormalities in DLBCL
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Diffuse Large B Cell Lymphoma, Gene Mutation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NGS Panel: patients who had NGS 481 gene mutation detected

INTERVENTIONS:
Other:

SUMMARY:
to detect the translocation of c-Myc, Bcl-2 and Bcl-6 by FISH and 481 gene mutation by next generation sequencing and analyze the relationship between this gene abnormalities and the efficacy and prognosis in diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
This is one arm, single center non-intervention study. New diagnosed diffuse large B cell lymphoma patients were enrolled to detect the translocation of c-Myc, Bcl-2 and Bcl-6 by FISH and 481 gene mutation by next generation sequencing, then patients received standard treatment with R-CHOP, R2CHOP and DA-EPOCH by investigate's choice according to the patients pathological characteristics. the basic characteristics and treatment response and progression-free survival and overall survival were collected and analyzed with the gene abnormalities. a total of 100 diffuse large B cell lymphoma patients will enrolled in one year and will finish after 3 years.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0-2;
* histological diagnosed diffuse large B cell lymphoma;
* normal hematological, hepatal, renal function;
* normal heart function with LVEF ≥ 50%;

Exclusion Criteria:

* Diagnosed as a malignant tumor other than lymphoma or receiving treatment, except for the following conditions:

  ①Have received treatment for the purpose of curing, and no malignant tumor with known active disease occurred ≥5 years before enrollment;

  ②Skin basal cell carcinoma (except melanoma) that has received adequate treatment and has no signs of disease;

  ③ Carcinoma in situ of the cervix that has received adequate treatment and has no signs of disease.
* Heart disease with clinical significance, including unstable angina pectoris, acute myocardial infarction within 6 months before screening.
* Congestive heart failure (NYHA) heart function is graded in grade III or IV (Annex 3)
* Severe arrhythmia requiring treatment.
* Patients with active hepatitis B and HIV infection.
* Women who are pregnant or breastfeeding
* Patients who have received organ transplants in the past
* Patients with severe active infection
* Have a history of severe neurological or psychiatric diseases, including dementia or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all new diagnosed DLBCL
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-02-08 (Estimated); Study Completion 2024-02-08 (Estimated)

PRIMARY OUTCOMES:
the incidence of gene mutation in DLBCL | 3 years
The incidence of gene mutation in different subtype of DLBCL | 3years
The relationship of ORR, progression free survival, overall survival of patients with standard treatment with gene abnormalities | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No